CLINICAL TRIAL: NCT07195383
Title: Evaluation of the Effects of Using the GUSS-ICU Safe Nutrition Program After Extubation in ICU Patients
Brief Title: GUSS-ICU Safe Nutrition Program After Extubation in ICU Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Zeliha Tülek, Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-74555795-050.04-1249240
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Dysphagia; Dysphagia, Swallowing Function, Diet Modification, Dysphagia Diet, Diet Standardization
Keywords: DYSPHAGIA; ICU; POST- EXTUBATION
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GUSS-ICU Applied Group (Experimental): The GUSS-ICU Scale, which is used for the transition to feeding of extubated patients, will be applied to the randomly selected intervention group included in the study, and feeding will be planned and continued for 4 days according to the score achieved.
  Interventions: Other: Nutrion plan based on GUSS-ICU scale
- Routine Follow-up Group (No Intervention): Routine care and follow-up will be applied to the randomly selected control group for 4 days after extubation.

INTERVENTIONS:
Other: Nutrion plan based on GUSS-ICU scale — To ensure a rapid and accurate transition to post-extubation nutrition, patients will be assessed using the GUSS-ICU scale at 4 hours after extubation. A nutrition plan will be created based on the patient's GUSS-ICU score and will be maintained for 4 days.
  Other Names: Use of the GUSS-ICU scale after extubation
  Arms: GUSS-ICU Applied Group

SUMMARY:
The aim of this study is to evaluate the effects of using the GUSS-ICU Safe Nutrition Program after extubation in Intensive Care Unit patients. This randomized controlled trial will be conducted in the Anesthesia Intensive Care Unit of Bakırköy Dr. Sadi Konuk Training and Research Hospital. Eligible participants will be randomly assigned to either the control group (usual care/routine follow-up group) or the intervention group (GUSS-ICU patients). Patients undergoing GUSS-ICU assessment will continue the nutritional program, as directed by the scale, for four days. Data are recorded on the first and last day. The data will then be evaluated in conjunction with the control group data.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effects of using the GUSS-ICU Safe Nutrition Program after extubation in intensive care patients. This randomized controlled trial will be conducted in the Anesthesia Intensive Care Unit of Bakırköy Dr. Sadi Konuk Training and Research Hospital. Patients who meet the criteria will be randomized into either an intervention group or a control group. Patients in the control group will receive routine post-extubation care, follow-up, and a nutrition plan. On day 1, baseline data will be collected using the m-NUTRIC score, APACHE-II, SOFA, Charlson Comorbidity Index (CCI), Scored Patient-Generated Subjective Global Assessment (PG-SGA), and a patient data form. Routine follow-up and nutrition plans will be continued. At the end of day 4, the m-NUTRIC score, APACHE-II, SOFA, Charlson Comorbidity Index (CCI), Scored Patient-Generated Subjective Global Assessment (PG-SGA), and a patient data form will be completed. Patients in the intervention group undergo a GUSS-ICU assessment within the first 4 hours after extubation. Nutrition planning is based on the assessment scores. On day 1, baseline data includes the m-NUTRIC score, APACHE-II, SOFA, Charlson Comorbidity Index (CCI), Scored Patient-Generated Subjective Global Assessment (PG-SGA), and a patient data form. Nutritional monitoring and follow-up are continued for 4 days. At the end of day 4, the m-NUTRIC score, APACHE-II, SOFA, Charlson Comorbidity Index (CCI), Scored Patient-Generated Subjective Global Assessment (PG-SGA), and a patient data form are completed. The data will then be evaluated in conjunction with the control group data.

ELIGIBILITY:
Inclusion Criteria:

Age 18 and over Patients expected to remain intubated for more than 24 hours. Patients who have been extubated for no more than 4 hours.

Exclusion Criteria:

* Patients with neuromuscular disease
* Patients requiring non-invasive ventilation for more than 6 hours after extubation
* Patients being followed in the terminal phase
* Patients with a tracheostomy cannula
* Patients with a history of dysphagia
* Patients with head/neck cancer or surgery
* Patients with existing facial fractures
* Patients with a RASS score not within the 0-2 range
* Patients at high risk of bleeding (INR ≥ 2.0, Platelet count ≤ 50,000).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in malnutrition risk scores and findings in intensive care patients who received a GUSS-ICU Safe Nutrition Program after extubation | On the 1st and 4th days after extubation
  Changes in malnutrition risk scores and findings in intensive care patients who received the GUSS-ICU Safe Nutrition Program after extubation will be evaluated with the PG-SGA.
Changes in dehydration findings in intensive care patients who received a GUSS-ICU Safe Nutrition Program after extubation | On the 1st and 4th days after extubation
  Dehydration findings in intensive care patients who are applied GUSS-ICU Safe Nutrition Program after extubation will be evaluated with PG-SGA and patient data form.
Change in the incidence of aspiration pneumonia in intensive care patients receiving a GUSS-ICU safe nutrition program after extubation | On the 1st and 4th days after extubation
  The data in the patient follow-up form will be evaluated with the clinician's supervision.
Change in the frequency of GI symptoms in intensive care patients who received a post-extubation GUSS-ICU safe nutrition program | On the 1st and 4th days after extubation
  Changes in the frequency of GI symptoms in intensive care patients who received a GUSS-ICU Safe Nutrition Program after extubation will be evaluated with PG-SGA and Patient Data Form.

SECONDARY OUTCOMES:
Change in Modified Nutrition Risk in the Critically Ill (m-NUTRIC) score | On the 1st and 4th days after extubation
  It will be assessed with the Modified Nutrition Risk in the Critically Ill (m-NUTRIC) score.
Change in APACHE II score | On the 1st and 4th days after extubation
  The effects on mortality will be evaluated with the APACHE II score.
Change in SOFA (Sequential Organ Failure Assessment) Score | On the 1st and 4th days after extubation
  SOFA (Sequential Organ Failure Assessment) Score will be evaluated to determine the effects on mortality.
Change in Scored Patient-Generated Subjective Global Assessment (PG-SGA) score | On the 1st and 4th days after extubation
  Possible effects on nutrition will be evaluated using the Scored Patient-Generated Subjective Global Assessment (PG-SGA).

OTHER OUTCOMES:
Change in the number of days from tube feeding to oral feeding | From the first to the last day of follow-up after extubation
  Change in the number of days from tube feeding to oral feeding
Change in oral intake (calorie) | From the first to the last day of follow-up after extubation
  Change in oral intake (calorie)

CONTACTS AND LOCATIONS:
Overall Officials: Merve TURKAY, Principal Investigator — Istanbul Universitesi-Cerrahpasa; Zeliha TÜLEK, Study Director — Istanbul Universitesi-Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul
  - Istanbul Universitesi-Cerrahpasa, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhuley JN, Naik SR. Moderate protective effect of 6-MFA, a microbial metabolite obtained from Aspergillus ochraceus on immunological liver injury in mice. Comp Immunol Microbiol Infect Dis. 1999 Jan;22(1):15-25. doi: 10.1016/s0147-9571(98)00021-6. PMID 10099025